CLINICAL TRIAL: NCT03966716
Title: HipSTHeR - a Registerbased Randomized Controlled Trial - Hip Screws or (Total) Hip Replacement for Undisplaced Femoral Neck Fractures in Elderly Patients.
Brief Title: Hips Screws or (Total) Hip Replacement for Undisplaced Femoral Neck Fractures in Elderly Patients (HipSTHeR)
Acronym: HipSTHeR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-00140
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Femoral Neck Fractures; Undisplaced Fracture
Keywords: Internal Fixation; Hip Arthroplasty; Reoperation Rate; Mortality; Health Economy; External validity; Adverse events
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Arthroplasty; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arthroplasty (Experimental): Arthroplasty, hemi or total depending on patient characteristics and surgeon's choice
  Interventions: Device: Arthroplasty
- Internal Fixation (Active Comparator): Internal fixation with 2-3 screws or pins, or sliding hip screw device, depending on each hospital's routine
  Interventions: Device: Internal Fixation

INTERVENTIONS:
Device: Arthroplasty — Patients with an undisplaced femoral neck fracture receive a hemi or total hip arthroplasty depending on each hospital's routine for patient age and mobility.
  Arms: Arthroplasty
Device: Internal Fixation — Patients with an undisplaced femoral neck fracture undergo a closed reduction and internal fixation with 2-3 screws or pins, or sliding hip screw device. Type of fixation depends on each hospital's routine.
  Arms: Internal Fixation

SUMMARY:
A registerbased RCT will investigate whether arthroplasty can decrease the reoperation rate compared to internal fixation for patients with an undisplaced femoral neck fracture (Garden I-II).

DETAILED DESCRIPTION:
The aim of this study is to determine whether the treatment of elderly patients with an undisplaced femoral neck fracture (uFNF) can be improved by decreasing reoperation rates through replacing the hip instead of trying to preserve it. Patients ≥75 years with an uFNF will be included and randomized within the Swedish Fracture Register (SFR) platform to internal fixation (screws/pins) or arthroplasty (choice of hemi or total is at the surgeon's discretion). The primary outcome will be a composite variable that combines two variables (reoperations and mortality) into a single variable.

ELIGIBILITY:
Inclusion Criteria:

* Undisplaced (Garden I-II) femoral neck fracture (within 72h)
* treated at participating unit
* informed consent
* amenable for both treatment options

Exclusion Criteria:

* no informed consent
* pathological or stress fracture
* peri-implant fracture

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Composite variable comprising reoperation rate and mortality | 1 to 2-year post-surgery
  Both Death and mortality will be accounted for

SECONDARY OUTCOMES:
Reoperation rate | 2-year post-surgery
  Minor and major reoperations will be noted
Long-term Mortality | 2-year post-surgery
  All deaths are recorded
Short-term Mortality | 30 day mortality
  All deaths are recorded
Patient reported outcome: SMFA | 1-year post surgery
  Short Musculoskeletal Functional Assessment (SMFA) questionnaire, will be routinely collected within the Swedish Fracture Register 1 year after the injury and compared with the results obtained by recall technique at the time of the fracture.

OTHER OUTCOMES:
Occurrence of adverse events. | 1-year post-surgery
  Adverse events, such as pulmonary embolism, infection, dislocation, myocardial infarction and stroke will be noted.
Long-term reoperation rate | 5 and 10 years post-surgery
  Minor and major reoperations will be noted
External validity | 2-year post-surgery
  Assessment of eligible patients not included in the study

CONTACTS AND LOCATIONS:
Overall Officials: Stergios Lazarinis, Study Chair — Uppsala University Hospital
Locations (25):
- Sweden (25):
  - Uppsala University Hospital, Uppsala, Uppsala County
  - Alingsås Hospital, Alingsås
  - Borås Hospital, Borås
  - Falu Hospital, Falun
  - Gävle Hospital, Gävle
  - Sahlgrenska university Hospital, Gothenburg
  - Jönköping Hospital, Jönköping
  - Kalmar Hospital, Kalmar
  - Karlskrona Hospital, Karlskrona
  - Kungälv Hospital, Kungälv
  - Linköping University Hospital, Linköping
  - Sunderby Hospital, Luleå
  - Lycksele Hospital, Lycksele
  - Skåne Universitetssjukhus, Malmo
  - Mora Hospital, Mora
  - Norrtälje Hospital, Norrtälje
  - Nyköping Hospital, Nyköping
  - Skellefteå Hospital, Skellefteå
  - Skövde Hospital, Skövde
  - Danderyd Hospital, Stockholm
  - Stockholm South Hospital, Stockholm
  - Trollhättan Hospital, Trollhättan
  - Umeå University Hospital, Umeå
  - Västerås Hospital, Västerås
  - Västervik Hospital, Västervik

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Onativia IJ, Slullitel PA, Diaz Dilernia F, Gonzales Viezcas JM, Vietto V, Ramkumar PN, Buttaro MA, Piuzzi NS. Outcomes of nondisplaced intracapsular femoral neck fractures with internal screw fixation in elderly patients: a systematic review. Hip Int. 2018 Jan;28(1):18-28. doi: 10.5301/hipint.5000532. PMID 28665454
- [Background] Dolatowski FC, Frihagen F, Bartels S, Opland V, Saltyte Benth J, Talsnes O, Hoelsbrekken SE, Utvag SE. Screw Fixation Versus Hemiarthroplasty for Nondisplaced Femoral Neck Fractures in Elderly Patients: A Multicenter Randomized Controlled Trial. J Bone Joint Surg Am. 2019 Jan 16;101(2):136-144. doi: 10.2106/JBJS.18.00316. PMID 30653043
- [Derived] Wolf O, Sjoholm P, Hailer NP, Moller M, Mukka S. Study protocol: HipSTHeR - a register-based randomised controlled trial - hip screws or (total) hip replacement for undisplaced femoral neck fractures in older patients. BMC Geriatr. 2020 Jan 21;20(1):19. doi: 10.1186/s12877-020-1418-2. PMID 31964340